CLINICAL TRIAL: NCT01326663
Title: A Double Blind Trial Of Divalproex Sodium For Affective Lability And Alcohol Use Following Traumatic Brain Injury
Brief Title: Divalproex Sodium for Mood Swings and Alcohol Use Following Head Injury.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Paul Saenger (Other)
Responsible Party: Sponsor-Investigator, Paul Saenger, Executive Director, Denver Research Institute
Organization: Denver Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT075168
Record Dates: First submitted 2011-03-29; First posted 2011-03-31 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Veterans; TBI; Alcoholism; Irritable Mood
Keywords: Veterans; TBI; Alcoholism; Mood
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- divalproex sodium (Active Comparator)
  Interventions: Drug: Medication Trial
- sugar pill (Placebo Comparator)
  Interventions: Drug: Medication Trial

INTERVENTIONS:
Drug: Medication Trial

SUMMARY:
Despite the body's natural healing during the first year after a head injury, many veterans who have suffered even mild brain injuries find themselves easily upset or fearful as they go about their daily lives. While these reactions to the world around them were easily managed before the head injury, they now occur with little or no interruption and are exceedingly difficult to manage. Such reactions include a sense of always being upset or fearful that often makes it difficult to get along with family members, friends, coworkers, and employers. This may lead to broken marriages, unemployment, and even homelessness.

Some people with head injuries try to manage their unmanageable moods by drinking alcohol because it can create a sense of calm. However, alcohol's actions are short in duration. Most find that they have to drink more and more for a similar calming effect, and they soon become dependent on alcohol. This makes working and being part of their families even more difficult.

To treat the unmanageable mood, we tried a medicine called valproate, one that eases mood problems in people without head injury. We gave valproate to head injured persons with mood problems in a "non-blinded" study where both the doctor and the patient knew that the medicine was valproate and both were optimistic that it would work. In a small sample of eighteen people, 85% found mood relief and most of those either stopped drinking alcohol or drank much less than before. However, this might have been because both the doctor and patient were hopeful that the medication would make the patient feel better or because the medicine actually worked.

The only way to know for sure if the medicine works is to perform a study in which people receive either valproate or a sugar pill while neither they nor their doctor know which one they are taking. This is called a double blind study, as proposed here, and will involve nearly three times as many head injured persons as the first study.

If it is successful, this study will show that valproate treatment helps head injured people manage their moods and allows them to return to families, friends, and work. It will also show that they drink alcohol less or not at all, improving their health even further. Then doctors will know that they can use this medicine for large numbers of people who suffer from head injury and help them to lead normal lives. If the outcome of the study shows that the medicine works well, doctors can then use this medicine to treat people with head injury immediately after the study results are published.

ELIGIBILITY:
Inclusion Criteria:

* a history of remote (≥ 1 year prior to study enrollment) non-penetrating TBI
* currently using alcohol
* symptoms of affective lability: mood swings, irritability, frustration

Exclusion Criteria:

* a history of bipolar disorder or anxiety disorder prior to any head injury
* a history of head injury in which the cranium was opened either traumatically or surgically
* a history of stroke
* a history of seizure disorder other than those caused by ethanol withdrawal
* evidence of active liver disease
* current diagnosis or past history of major psychosis, the alcohol amnesic syndrome, or any type of dementia
* current suicidal/homicidal ideations
* any medical conditions that would constitute contraindications to treatment with divalproex sodium
* currently taking any medications that are known to affect the metabolism of divalproex sodium

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-10; Primary Completion 2013-05 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Reduced Affective Lability | Study weeks 1-10
  The primary analysis addresses our primary hypothesis that treatment with divalproex sodium will lessen affective lability significantly (p<0.05) as compared to placebo. We will characterize affective lability using discrete variables of presence or extent of symptoms yielded by the Neurobehavioral Rating Scale-Revised (Levin et al., 1990) as well as eight target items from the Agitated Behavior Scale (Bogner et al., 2000). Average intensity and duration of affective lability will be compared between groups.

SECONDARY OUTCOMES:
Reduced Alcohol Use | Study weeks 1-10
  The secondary analysis first addresses our secondary hypothesis that treatment with divalproex sodium will lessen quantity and frequency of ethanol use significantly (p<0.05) as compared to placebo in a sample of TBI subjects. We will characterize drinking using the Time Line Follow-Back for Drugs and Alcohol method, developed by Sobell et al (Sobell et al., 1979).

CONTACTS AND LOCATIONS:
Locations (1):
- Denver Veteran's Affairs Medical Center, Denver, Colorado, United States